CLINICAL TRIAL: NCT06420791
Title: The Dual Impact of Cirrhosis on Transplantation for Hepatocellular Carcinoma：a Two-center Retrospective Cohort Study in China
Status: Completed | Type: Observational
Sponsor: Xiao Xu (Other)
Responsible Party: Sponsor-Investigator, Xiao Xu, Principal Investigator, Clinical Professor,PHD,MD, Zhejiang University
Organization: Zhejiang University (Other)
Other Study IDs: CT2024-ZJU-OBS9
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
Background: This study aims to investigate the correlation between cirrhosis and hepatocellular carcinoma (HCC) recurrence after Liver Transplantation.

Methods: The study retrospectively collected data enrolled from 519 HCC patients who underwent liver transplantation from two center(the First Affiliated Hospital, Zhejiang University School of Medicine and Shulan (Hangzhou) Hospital, January 2015 to December 2020), Based on important variables, 1:3 propensity score matching (PSM) were performed respectively.

ELIGIBILITY:
Inclusion Criteria:

The patients undergoing liver transplantation for HCC from January 2015 to December 2020.

Exclusion Criteria:

Re-transplantation or combined liver-kidney transplantation; incomplete laboratory or clinical data; death within 90 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously registered liver transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
The overall survival rate was evaluated by follow-up investigation and outpatient review | 2-5 years

SECONDARY OUTCOMES:
The tumor-free survival rate was evaluated by follow-up investigation and outpatient review | 2-5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University school of Medicine, Hangzhou, Zhejiang, China